CLINICAL TRIAL: NCT06995287
Title: Evaluation of the Analgesic Effect of Intramyometrial Botulinum Toxin Injection Via Hysteroscopy in Severe Primary Dysmenorrhea: a Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Evaluation of the Analgesic Effect of Intramyometrial Botulinum Toxin Injection Via Hysteroscopy in Severe Primary Dysmenorrhea
Acronym: HYSTEROXINE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC24_0428; 2025-520638-53-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Dysmenorrhea; Chronic Pelvic Pain
Keywords: Primary dysmenorrhea; injection; Botulimum toxin, Type A
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A (Experimental): One injection will be performed via hysteroscopy under local anesthesia. The patient will be followed up remotely at M1 and M6 to complete questionnaires, and will be seen in site at M3 for a postoperative consultation and to complete questionnaires.
  Interventions: Drug: Xeomin
- Placebo (Placebo Comparator): One injection will be performed via hysteroscopy under local anesthesia. The patient will be followed up remotely at M1 and M6 to complete questionnaires, and will be seen in site at M3 for a postoperative consultation and to complete questionnaires.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xeomin — One injection will be performed via hysteroscopy under local anesthesia.
  Arms: Botulinum toxin type A
Drug: Placebo — One injection will be performed via hysteroscopy under local anesthesia.
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the global impression of improvement at 3 months following intramyometrial botulinum toxin injections via hysteroscopy in women with severe primary dysmenorrhea who have failed first-line medical treatment, compared to intramyometrial placebo injections.

DETAILED DESCRIPTION:
This trial is multicenter, placebo-controlled, randomized with center-based stratification, double-blind and prospective. The treatment consists of a single injection follow by 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult women who are not menopausal,
* Experiencing severe dysmenorrhea, defined as an average pain intensity score ≥ 6/10 on a Numerical Rating Scale (NRS) over the past 3 months at the inclusion visit,
* Having failed optimal first-line medical treatment combining hormonal therapy and appropriate analgesics (Level I and II analgesics, and NSAIDs),
* Having undergone a pelvic MRI within 6 months prior to the inclusion visit that shows no evidence of deep infiltrating endometriosis or endometrioma, following systematic review by radiologists from the expert center managing the patient (if the pelvic MRI is deemed of insufficient quality for interpretation, a new MRI will be performed at the center),
* Using a highly effective method of contraception (failure rate <1%) for the entire duration of the follow-up period. Highly effective contraception methods are defined as one of the following: combined hormonal contraception (containing estrogen and progestin) with ovulation inhibition (oral, vaginal, or transdermal), progestin-only hormonal contraception with ovulation inhibition (oral, injectable, or implantable), intrauterine device (IUD), intrauterine hormonal system (IUS), condoms, bilateral tubal occlusion, vasectomized partner, or sexual abstinence,
* Having a negative urine pregnancy test on the day of the procedure,
* Having signed the informed consent form for the study at the M-1 visit.

Exclusion Criteria:

* Pregnant or planning a pregnancy during the entire study period,
* Currently breastfeeding,
* Refusal to use effective contraception during the study and for 6 months after its completion,
* Contraindications to botulinum toxin, including:
* Generalized disorders of muscular activity (e.g., myasthenia gravis, Lambert-Eaton syndrome),
* Ongoing treatment with aminoglycosides, peripheral muscle relaxants, or amino-4-quinolines,
* Hypersensitivity to the active substance, human albumin, or sucrose,
* Bleeding disorders or current treatment with anticoagulants,
* Ongoing vaginal or upper genital tract infection,
* Participation in another interventional clinical trial,
* Inability to cooperate or understand the study requirements in a way that would allow strict adherence to the protocol,
* Subject to legal protection measures (e.g., guardianship, curatorship, or judicial protection),
* Not affiliated with the French social security system,
* Unable to access the internet to complete questionnaires at Month 1 and Month 6.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2026-02-09 (Actual); Primary Completion 2028-06-09 (Estimated); Study Completion 2028-09-09 (Estimated)

PRIMARY OUTCOMES:
Patient Global Improvement | 3 months
  The response (favorable versus unfavorable) to the Patient Global Impression of Improvement questionnaire at 3 months following intra-myometrial injection. A response is considered favorable when the score of Patient Global Impression of Improvement questionnaire is 1 or 2. Patient Global Impression of Improvement questionnaire is self-assessment scale ranging from 1 (Very much improved) to 7 (Very much worsened).

SECONDARY OUTCOMES:
Average intensity of dysmenorrhea | 6 months
  Average intensity of dysmenorrhea evaluated using a numerical rating scale during the last menstrual cycle before injection, then at 3 and 6 months. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Maximum intensity of dysmenorrhea | 6 months
  Maximum intensity of dysmenorrhea evaluated using a numerical rating scale during the last menstrual cycle before injection, then at 3 and 6 months. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Duration of dysmenorrhea | 6 months
  Duration (in days) of dysmenorrhea during the last menstrual cycle before injection, then at 3 and 6 months.
Average intensity of non-menstrual pelvic pain | 6 months
  Average intensity of non-menstrual pelvic pain evaluated using an numerical rating scale before injection, then at 1, 3, and 6 months. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Maximum intensity of non-menstrual pelvic pain | 6 months
  Maximum intensity of non-menstrual pelvic pain evaluated using an numerical rating scale before injection, then at 1, 3, and 6 months. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Duration of non-menstrual pelvic pain | 6 months
  Duration of non-menstrual pelvic pain (in days) evaluated before injection, then at 1, 3, and 6 months
Average intensity of pain during the most recent sexual intercourse | 6 months
  Average intensity of pain during the most recent sexual intercourse, evaluated using an numerical rating scale before injection, then at 1, 3, and 6 months. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Sexual function assessed using the Female Sexual Function Index | 6 months
  Sexual function assessed using the Female Sexual Function Index before injection, and then at 1, 3, and 6 months. The Female Sexual Function Index consists of 19 items assessing six dimensions of female sexual function (desire, arousal, pain, lubrication, satisfaction, orgasm). The total score ranges from 2 to 36, with sexual dysfunction defined as a score below 23.
Central sensitization to pain | 3 months
  Central sensitization to pain assessed using the Convergences PP score, before injection and at 3 months. The total Convergence PP score ranges from 0 to 10, with pelvic hypersensitivity defined as a score greater than or equal to 5.
Heavy menstrual bleeding assessed using the Higham score | 6 months
  Heavy menstrual bleeding assessed using the Higham score during the last menstrual period, before injection, and at 3 and 6 months. The Higham score is an objective assessment score of menstrual blood loss. Each day of menstruation, the patiente counts the number of pads or tampons used, referring to a visual chart. A score above 100 points corresponds to a blood loss of 80 mL, which defines menorrhagia.
General quality of life | 6 months
  General quality of life assessed using the The Short Form (36) Health Survey before injection, and at 1, 3, and 6 months. The questionnaire The Short Form (36) Health Survey is a multidimensional, generic scale, meaning it assesses health status regardless of the underlying condition, gender, age, or treatment. Its 36 items evaluate 8 domains: physical activity, physical role limitations, bodily pain, perceived health, vitality, social functioning, emotional state, and mental health. Each item is scored from 0 (lowest score) to 100 (highest score). At the end, a score for each SF-36 dimension is calculated based on the corresponding items, ranging from 0 (poor quality of life) to 100 (best quality of life).
Disease-specific quality of life | 6 months
  Disease-specific quality of life assessed using the Endometriosis Health Profile EHP-5 questionnaire (it is the short version of Endometriosis Health Profile EHP-30) before injection, and at 1, 3, and 6 months. This short questionnaire includes only 11 out of 30 questions, to which patients must respond with Always, Often, Sometimes, Rarely, or Never. This questionnaire ranging from 0 (the best health status) to 44 (the worst health status).
Number of days of school or work absenteeism | 6 months
  Number of days of school or work absenteeism in the past month, assessed before injection and at 1, 3, and 6 months.
Anxiety assessed using the State and Tait Anxiety Inventoy-Y scale | 3 months
  Anxiety assessed using the State and Tait Anxiety Inventoy scale-Y before injection and at 3 months. This State and Tait Anxiety Inventoy scale-Y includes two distinct scales for assessing state anxiety (STAI Form Y-A) and trait anxiety (STAI Form Y-B). The Trait Anxiety scale consists of 20 items and assesses the individual's general tendency to experience anxiety. Scores range from 21 to 77.
  The State Anxiety scale also includes 20 items and measures a temporary anxious mood (stress). Scores range from 20 to 80.
Depression evaluated using the Beck Depression Inventory-II | 3 months
  Depression evaluated using the Beck Depression Inventory-II before injection and at 3 months. This is a self-administered questionnaire consisting of 21 items. Each item includes 4 statements corresponding to increasing levels of symptom intensity, rated on a scale from 0 to 3. The total score is obtained by summing the scores of the 21 items. The score can be interpreted according to the following four categories: no depression (score < 10); mild depression (10 < score < 18); moderate depression (19 < score < 29); and severe depression (score > 30).
Global improvement percentage | 6 months
  Global improvement percentage (0-100%) assessed at 1, 3, and 6 months.
Pain intensity during the procedure | during procedure
  Pain intensity during the procedure assessed via numerical rating scale. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Pain intensity at 5 minutes post-procedure | 5 minutes post-procedure
  Pain intensity at 5 minutes post-procedure, assessed via numerical rating scale
Adverse events related to the injections | 6 months
  Adverse events related to the injections, recorded immediately postoperatively, and at 1, 3, and 6 months.
Emergency visits following the procedure | 1 month
  Emergency visits following the procedure, assessed at 1 month.
Exploratory analysis for the MEOPA subgroup : Primary Outcome | 3 months
  Exploratory analysis for the MEOPA subgroup: Primary outcome. The response (favorable versus unfavorable) to the Patient Global Impression of Improvement questionnaire at 3 months following intra-myometrial injection. A response is considered favorable when the score of Patient Global Impression of Improvement questionnaire is 1 or 2. Patient Global Impression of Improvement questionnaire is self-assessment scale ranging from 1 (Very much improved) to 7 (Very much worsened).
Exploratory analysis for the MEOPA subgroup : Pain intensity during the procedure | during procedure
  Exploratory analysis for the MEOPA subgroup : procedural pain. Pain intensity during the procedure assessed via numerical rating scale. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Exploratory analysis for the MEOPA subgroup: Willingness to repeat the intervention | 6 months
  Exploratory analysis for the MEOPA subgroup: willingness to repeat the intervention. The response is rating Yes or No.
Exploratory analysis for the MEOPA subgroup: Adverse event | 6 months
  Exploratory analysis for the MEOPA subgroup: adverse events.
Exploratory analysis for the MEOPA subgroup : Emergency visits | 6 months
  Exploratory analysis for the MEOPA subgroup : emergency visits.
Exploratory analysis for the hormonal treatment subgroup : Primary Outcome | 3 months
  Exploratory analysis for the hormonal treatment subgroup : Primary outcome. The response (favorable versus unfavorable) to the Patient Global Impression of Improvement questionnaire at 3 months following intra-myometrial injection. A response is considered favorable when the score of Patient Global Impression of Improvement questionnaire is 1 or 2. Patient Global Impression of Improvement questionnaire is self-assessment scale ranging from 1 (Very much improved) to 7 (Very much worsened).
Exploratory analysis for the hormonal treatment subgroup : Pain intensity during the procedure | during procedure
  Exploratory analysis for the hormonal treatment subgroup : procedural pain. Pain intensity during the procedure assessed via numerical rating scale. Numerical rating scale is self-assessment scale ranging from 0 (no pain) to 10 (maximum imaginable pain).
Exploratory analysis for the hormonal treatment subgroup : Willingness to repeat the intervention | 6 months
  Exploratory analysis for the hormonal treatment subgroup : willingness to repeat the intervention. The response is rating Yes or No.
Exploratory analysis for the hormonal treatment subgroup : Adverse event | 6 months
  Exploratory analysis for the hormonal treatment subgroup : adverse events.
Exploratory analysis for the hormonal treatment subgroup : Emergency visits | 6 months
  Exploratory analysis for the hormonal treatment subgroup : emergency visits.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Clinique axium / Centre resilience, Aix-en-Provence
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU Lille, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - CHU Nantes, Nantes
  - Clinique Brétéché, Nantes
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided